CLINICAL TRIAL: NCT01657214
Title: Phase I, Dose Escalation Study of Safety, Pharmacokinetic and Pharmacodynamic of SAR125844 Administered Weekly as Intravenous Infusion in Asian Adult Patients With Advanced Malignant Solid Tumors
Brief Title: Phase I, Dose Escalation of SAR125844 in Asian Solid Tumor Patients
Acronym: SARMETA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED12337; U1111-1126-7527 (Other: UTN)
Record Dates: First submitted 2012-07-24; First posted 2012-08-06 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — SAR125844

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): SAR125844 will be administered as weekly IV infusion. Four weekly administrations are considered as 1 cycle. The starting dose will be either 1 dose level (DL) below the highest cleared dose level in a European TED11449 ongoing study or DL4 (260 mg/m^2), if the highest cleared dose in TED11449 is >340 mg/m^2.
  Interventions: Drug: SAR125844

INTERVENTIONS:
Drug: SAR125844 — Pharmaceutical form:Concentrate for solution
  Route of administration: intravenous

SUMMARY:
Primary Objective:

In the dose escalation: to determine the maximum tolerated dose (MTD) of SAR125844.

In the expansion cohort: to evaluate the preliminary anti-tumoral effect of SAR125844 in patients with measurable and MET gene amplification (including gastric cancer patients).

Secondary Objectives:

To characterize and confirm the global safety profile of SAR125844 including cumulative toxicities.

To assess preliminary antitumor activity of SAR125844. To explore the pharmacodynamic effects (PDy) of SAR125844. To evaluate the pharmacokinetic profile of SAR125844. To explore the relationship of MET gene amplification status with antitumor effects.

To evaluate other pharmacodynamic biomarkers.

DETAILED DESCRIPTION:
For both cohorts, escalation and expansion, the duration of the study for one patient will include a period for inclusion of up to 3 weeks and a 4-week treatment cycle(s).The patient may continue treatment until disease progression, unacceptable toxicity or willingness to stop, followed by a minimum of 30-days follow-up.

If a patient treated in dose escalation part or in an expansion cohort, continues to benefit from the treatment at the time of Clinical Study Report, the patient can continue study treatment for a maximum of 1 year and will continue to undergo all assessments as per the study flowchart. Such patients will be followed at least until 30 days after the last IMP administration.

ELIGIBILITY:
Inclusion criteria:

* Patients with solid tumor for which no standard therapy is available.
* At the recommended dose (expansion cohort): only patients with measurable disease and MET gene amplification.

Exclusion criteria:

* Patient less than 20 years old.
* ECOG performance status >2.
* Poor bone marrow reserve as defined by absolute neutrophils count <1.5 x 10^9/L or platelets <100 x 10^9/L.
* Poor organ function as defined by one of the following:
* Total bilirubin >1.5 x ULN.
* AST, ALT, alkaline phosphatase >2.5 x ULN or >5 x ULN in case of documented liver metastasis.
* Serum creatinine >1.5 x ULN, or serum creatinine between 1.0 and 1.5 x ULN associated with calculated creatinine clearance <60 mL/min.
* Proteinuria >500mg/24h.
* Pregnant or breast-feeding women.
* Sexually active (males and females) who do not agree to use medically acceptable methods of contraception during the course of the study and for 3 months following discontinuation of study drug.
* Female patients of childbearing potential must have a negative pregnancy test at screening.
* Known or symptomatic brain metastasis (other than totally resected or previously pre-irradiated and no progressive/relapsing) or lepto-meningeal carcinomatosis.
* No resolution of any specific toxicities (excluding alopecia) related to any prior anti-cancer therapy to grade ≤1 according to the NCI CTCAE v.4.03.
* Wash out period of less than 3 weeks from previous antitumor therapy or any investigational treatment,(and less than 6 weeks in case of prior nitrozo-urea and or mitomycin C treatment).
* Any surgery with major risk of bleeding performed less than 10 days prior to study treatment administration.
* Any other severe underlying medical conditions, which could impair the ability to participate in the study.
* Patients treated with potent CYP3A inhibitor.
* Patients treated with potent and moderate CYP3A inducers.
* Known hypersensitivity or any adverse event related to the study drug excipient (Captisol®).
* Prior treatment with any MET inhibitor compound (selective or not).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
- DOSE ESCALATION To determine the maximum tolerated dose (MTD) of SAR125844 | At d28 of Cycle 1 of each treated patient, DLT is assessed
- EXPANSION Cohort To evaluate the preliminary anti-tumoral effect of SAR125844 | Antitumor activity is assessed at the end of Cycle 1, then every 2 cycles up to treatment discontinuation

SECONDARY OUTCOMES:
Number of patients with treatment emergent events | Up to a maximum of 2 years
Assessment of PK parameter Cmax | Up to a maximum of 2 years
Assessment of PK parameter AUCs | Up to a maximum of 2 years
Assessment of PK parameter CL | Up to a maximum of 2 years
Assessment of PD parameter ShedMET | Up to a maximum of 2 years
Assessment of PD parameter HGF | Up to a maximum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Japan (4):
  - Investigational Site Number 392001, Kashiwa-Shi
  - Investigational Site Number 392004, Suita-Shi
  - Investigational Site Number 392002, Sunto-Gun
  - Investigational Site Number 392003, Takatsuki-Shi
- South Korea (4):
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410002, Seoul